CLINICAL TRIAL: NCT00535626
Title: A Post-market, Non-randomized, Open Label, Multi-center Clinical Study of the Trident Tritanium Acetabular Shell
Brief Title: Trident® Tritanium™ Acetabular Shell Revision Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 61
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trident® Tritanium™ Acetabular Shell (Other): Trident® Tritanium™ Acetabular Shell used in revision total hip replacement
  Interventions: Device: Trident® Tritanium™ Acetabular Shell

INTERVENTIONS:
Device: Trident® Tritanium™ Acetabular Shell — Trident® Tritanium™ Acetabular Shell

SUMMARY:
The purpose of this study is to evaluate a hip implant system used when a previous hip replacement surgery has failed.

DETAILED DESCRIPTION:
Total hip replacement is considered to be a very successful surgical procedure for the treatment of degenerative joint disease. Clinical results for cementless acetabular components have demonstrated excellent long-term fixation of these devices. However, so called 'first generation' cementless acetabular components have not had similar success rates. In these cases the acetabular component is often revised due to loosening, wear or infection.

Revision hip arthroplasty also becomes a challenge as patients often present with severe bone loss and poor bone quality. This can lead to compromised initial stability, which in turn leads to lack of long-term fixation and failure. Acetabular revision with a cementless component has shown improved results over cemented fixation.

Radiographic evaluation of the Trident® Tritanium™ Acetabular Shell will provide valuable early to intermediate information that may help predict the long-term success of this new system.

It is the intention of this study to closely follow subjects that have undergone revision hip replacement with regard to implant survivorship, signs of radiographic loosening, subjects' function evaluated through Harris Hip Score and Lower Extremity Activity Scale, subject quality of life through SF-36 and adverse events.

The primary efficacy hypothesis is that the rate of revision or pending revision (as defined by radiographic parameters) due to instability or lack of fixation for the Trident® Tritanium™ Acetabular Shell will be less than 10% at 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females, 21-85 years of age at the time of surgery.
2. Patient is a candidate for a revision of a failed acetabular component with a cementless acetabular component.
3. Patient has signed an IRB approved study consent form.
4. Patient is willing and able to comply with postoperative requirements including postoperative weight bearing restrictions and self-evaluations.

Exclusion Criteria:

1. Patient is morbidly obese, BMI > 40.
2. Patient has a systemic or metabolic bone disorder leading to progressive bone deterioration.
3. Patient is immunologically compromised or receiving steroids in excess of normal physiological requirements (> 30 days).
4. Patient's bone stock is compromised by disease or infection which cannot provide adequate support and/or fixation to the prosthesis.
5. Patient has an active or suspected latent infection on or about the hip joint.
6. Patient is a prisoner.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2006-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Malkani, MD, Study Chair — University of Louisville; Michael Masini, MD, Principal Investigator — St Joseph Mercy Hospital; Daniel Ward, MD, Principal Investigator — New England Baptist Hospital; Benjamin Bierbaum, MD, Principal Investigator — New England Baptist Hospital; Kirby Hitt, MD, Principal Investigator — Scott & White Memorial Hospital; Kenneth Greene, MD, Principal Investigator — Crystal Clinic; Jim Kudrna, MD, Principal Investigator — Illinois Bone & Joint Institute; Ivan Tomek, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Stephen Kantor, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Steven Barnett, MD, Principal Investigator — Orthopedic Specialty Institute; Carlos Higuera, MD, Principal Investigator — The Cleveland Clinic; Joseph Zuckerman, MD, Principal Investigator — NYU Hospital for Joint Diseases; Fredrick Jaffe, MD, Principal Investigator — NYU Hospital for Joint Diseases; Stephen Incavo, MD, Principal Investigator — The Methodist Hospital Research Institute; Timothy Lovell, MD, Principal Investigator — Rockwood Clinic; Sean Scully, MD, Principal Investigator — Cedars Medical Center; Amar Ranawat, MD, Principal Investigator — Hospital for Special Surgery, New York; Geoffrey Westrich, MD, Principal Investigator — Hospital for Special Surgery, New York; R D Heekin, MD, Principal Investigator — Heekin Institute for Orthopedic Research, Inc.; Bryce Allen, MD, Principal Investigator — Scott & White Memorial Hospital
Locations (15):
- United States (15):
  - Orthopedic Specialty Institute, Orange, California
  - Heekin Institute for Orthopedic Research, Inc., Jacksonville, Florida
  - Cedars Medical Center, Miami, Florida
  - Illinois Bone & Joint Institute, Glenview, Illinois
  - University of Louisville, 201 Abraham Flexner Way, Suite 100, Louisville, Kentucky
  - New England Baptist Hospital, Boston, Massachusetts
  - St Joseph Mercy Hospital, Ypsilanti, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Hospital for Joint Diseases, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Crystal Clinic, Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Methodist Hospital, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Rockwood Clinic, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 241 patients/245 hips - 51 patients/52 hips censored = 190 patients/193 hips followed
Units Other Than Participants: Hips
Period: Overall Study
Arm/Group | Trident® Tritanium™ Acetabular Shell
Started | 190; 193 Hips
Completed | 85; 86 Hips
Not Completed | 105; 107 Hips
Not completed — Death | 15
Not completed — Lost to Follow-up | 29
Not completed — Withdrawal by Subject | 20
Not completed — Removal/revision of study component | 8
Not completed — Subject terminated | 31
Not completed — Unable to return | 2

BASELINE CHARACTERISTICS:
Population: Participants who were not censored from analysis
Arm/Group | Trident® Tritanium™ Acetabular Shell
Number analyzed (Participants) | 190
Age, Continuous [Mean (Standard Deviation); unit: years] — For bilateral hip patients, the age at time of first study surgery is used.
  years | 63.70 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 105
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 190

OUTCOME MEASURES:

1. Primary Outcome: Number of Hips Requiring Revision or Pending Revision of the Acetabular Shell (as Defined by Radiographic Parameters) Due to Instability or Lack of Fixation
Time Frame: 5 years post-operative
Population: No cases were pending revision.
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | Trident® Tritanium™ Acetabular Shell
Number analyzed (Participants) | 190
Number analyzed (hips) | 193
hips | 4
Statistical Analysis 1: Comparison: Trident® Tritanium™ Acetabular Shell; Test type: Other — To test if revision rate at 5 years is less than 10% (Ha - Alternative Hypothesis). Note: All cases enrolled in the study had to undergo revision whether from their primary procedure or a previous revision. Based on literature, 10% is the expected rate of another revision occurring in this cohort of enrolled patients; Revision or Pending Revision Rate = 2.43, 90% CI 2-sided [1.07 to 5.46] — The estimated 2.43% revision rate was obtained by the Kaplan-Meier method

2. Secondary Outcome: Change in Harris Hip Score (HHS) From Pre-operative to Post-operative Visits
Description: The change in HHS is reported by comparing the mean pre-operative, 3-month, 1, 2, 3, 4, and 5 year post-operative scores. Scores can range from 0 to 100, with 0 being the worst and 100 being the best score. 90-100 = excellent, 80-89 = good, 70-79 = fair, 0-69 = poor.
Time Frame: pre-op, 3 month, 1, 2, 3, 4, 5 years
Population: Participants/hips with available data. Overall number of participants and units analyzed is based upon the preoperative population.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: hips
Arm/Group | Trident® Tritanium™ Acetabular Shell
Number analyzed (Participants) | 171
Number analyzed (hips) | 173
units on a scale
  Mean HHS score preoperative | 53.40 (21.99)
  Mean HHS score 3 months: number analyzed (Participants) | 147
  Mean HHS score 3 months: number analyzed (hips) | 149
  Mean HHS score 3 months | 79.46 (16.58)
  Mean HHS score 1 year: number analyzed (Participants) | 131
  Mean HHS score 1 year: number analyzed (hips) | 133
  Mean HHS score 1 year | 86.11 (14.83)
  Mean HHS score 2 years: number analyzed (Participants) | 116
  Mean HHS score 2 years: number analyzed (hips) | 117
  Mean HHS score 2 years | 85.34 (15.60)
  Mean HHS score 3 years: number analyzed (Participants) | 93
  Mean HHS score 3 years: number analyzed (hips) | 93
  Mean HHS score 3 years | 86.56 (15.40)
  Mean HHS score 4 years: number analyzed (Participants) | 83
  Mean HHS score 4 years: number analyzed (hips) | 83
  Mean HHS score 4 years | 83.87 (17.32)
  Mean HHS score 5 years: number analyzed (Participants) | 68
  Mean HHS score 5 years: number analyzed (hips) | 68
  Mean HHS score 5 years | 86.29 (14.43)
Statistical Analysis 1: Comparison: Trident® Tritanium™ Acetabular Shell; Test type: Other — To test if the change from the pre-operative HHS compared to the post-operative HHS at all intervals is statistically significant; p < 0.0001, t-test, 2 sided — This p-value applies to all intervals; Paired t-test

3. Secondary Outcome: Change in SF-36 From Pre-operative to Post-operative Visits
Description: The change in SF-36 is reported by comparing the mean preoperative, 3 month, 1, 2, 3, 4, and 5 year scores. The SF-36 Health Survey is a 36 item patient-completed questionnaire to measure general health and well-being. It includes a physical and mental status component score; each ranging from 0-100. Low values represent a poor health state and high values represent a good health state.
Time Frame: pre-op, 3 month, 1, 2, 3, 4, 5 years
Population: Participants/hips with available data. Overall number of participants and hips analyzed is based upon the preoperative population.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: hips
Arm/Group | Trident® Tritanium™ Acetabular Shell
Number analyzed (Participants) | 181
Number analyzed (hips) | 184
units on a scale
  Physical score preoperative | 33.26 (10.36)
  Physical score 3 months: number analyzed (Participants) | 160
  Physical score 3 months: number analyzed (hips) | 162
  Physical score 3 months | 38.9 (10.7)
  Physical score 1 year: number analyzed (Participants) | 143
  Physical score 1 year: number analyzed (hips) | 145
  Physical score 1 year | 43.04 (10.31)
  Physical score 2 years: number analyzed (Participants) | 121
  Physical score 2 years: number analyzed (hips) | 122
  Physical score 2 years | 43.55 (10.7)
  Physical score 3 years: number analyzed (Participants) | 104
  Physical score 3 years: number analyzed (hips) | 105
  Physical score 3 years | 43.54 (10.29)
  Physical score 4 years: number analyzed (Participants) | 99
  Physical score 4 years: number analyzed (hips) | 100
  Physical score 4 years | 42.76 (11.27)
  Physical score 5 years: number analyzed (Participants) | 79
  Physical score 5 years: number analyzed (hips) | 80
  Physical score 5 years | 43.82 (11.4)
  Mental score preoperative | 49.56 (13.08)
  Mental score 3 months: number analyzed (Participants) | 160
  Mental score 3 months: number analyzed (hips) | 162
  Mental score 3 months | 52.07 (11.4)
  Mental score 1 year: number analyzed (Participants) | 143
  Mental score 1 year: number analyzed (hips) | 145
  Mental score 1 year | 52.81 (10.44)
  Mental score 2 years: number analyzed (Participants) | 121
  Mental score 2 years: number analyzed (hips) | 122
  Mental score 2 years | 53.37 (10.22)
  Mental score 3 years: number analyzed (Participants) | 104
  Mental score 3 years: number analyzed (hips) | 105
  Mental score 3 years | 53.84 (9.67)
  Mental score 4 years: number analyzed (Participants) | 99
  Mental score 4 years: number analyzed (hips) | 100
  Mental score 4 years | 53.63 (10.29)
  Mental score 5 years: number analyzed (Participants) | 79
  Mental score 5 years: number analyzed (hips) | 80
  Mental score 5 years | 52.93 (9.25)
Statistical Analysis 1: Comparison: Trident® Tritanium™ Acetabular Shell; Test type: Other — To test whether the change from the pre-operative SF-36 Physical Score compared to each post-operative SF-36 Physical score is statistically significant; p < 0.0001, t-test, 2 sided — This p-value applies to all intervals; Paired t-test
Statistical Analysis 2: Comparison: Trident® Tritanium™ Acetabular Shell; Test type: Other — To test whether the change from the pre-operative SF-36 Mental Score compared to the 3 month SF-36 Mental Score is statistically significant; p = 0.0139, t-test, 2 sided; Paired t-test
Statistical Analysis 3: Comparison: Trident® Tritanium™ Acetabular Shell; Test type: Other — To test whether the change from the pre-operative SF-36 Mental Score compared to the 1 year SF-36 Mental Score is statistically significant; p = 0.0254, t-test, 2 sided; Paired t-test
Statistical Analysis 4: Comparison: Trident® Tritanium™ Acetabular Shell; Test type: Other — To test whether the change from the SF-36 Mental Score compared to the 2 year SF-36 Mental Score is statistically significant; p = 0.1506, t-test, 2 sided; Paired t-test
Statistical Analysis 5: Comparison: Trident® Tritanium™ Acetabular Shell; Test type: Other — To test whether the change from the pre-operative SF-36 Mental Score compared to the 3 year SF-36 Mental Score is statistically significant; p = 0.0936, t-test, 2 sided; Paired t-test
Statistical Analysis 6: Comparison: Trident® Tritanium™ Acetabular Shell; Test type: Other — To test if the change from the pre-operative SF-36 Mental Score compared to the 4 year SF-36 Mental Score is statistically significant; p = 0.0909, t-test, 2 sided; Paired t-test
Statistical Analysis 7: Comparison: Trident® Tritanium™ Acetabular Shell; Test type: Other — To test whether the change from the pre-operative SF-36 Mental Score compared to the 5 year SF-36 Mental Score is statistically significant; p = 0.048, t-test, 2 sided; Paired t-test

4. Secondary Outcome: Radiographic Outcomes: Radiolucency (RLL) Around the Acetabular Shell is Greater Than 2 mm in All Zones
Description: Defined as a lucent area seen parallel and in close proximity to the device at the prosthesis/bone interface encompassing at least 50% of the zone, and at least 1 mm or greater in width. May be accompanied by a radiopaque (reactive) line. Assessed for each of the three modified DeLee Charnley zones.
Time Frame: 3 month, 1, 2, 3, 4, 5 years
Population: Participants/hips are based on evaluable films for this data point. Overall number of participants and hips analyzed is based upon the 3 month population.
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | Trident® Tritanium™ Acetabular Shell
Number analyzed (Participants) | 152
Number analyzed (hips) | 154
hips
  RLL> 2mm in all zones at 3 months | 3
  RLL> 2mm in all zones at 1 year: number analyzed (Participants) | 133
  RLL> 2mm in all zones at 1 year: number analyzed (hips) | 135
  RLL> 2mm in all zones at 1 year | 0
  RLL> 2mm in all zones at 2 years: number analyzed (Participants) | 117
  RLL> 2mm in all zones at 2 years: number analyzed (hips) | 118
  RLL> 2mm in all zones at 2 years | 0
  RLL> 2mm in all zones at 3 years: number analyzed (Participants) | 90
  RLL> 2mm in all zones at 3 years: number analyzed (hips) | 90
  RLL> 2mm in all zones at 3 years | 0
  RLL> 2mm in all zones at 4 years: number analyzed (Participants) | 87
  RLL> 2mm in all zones at 4 years: number analyzed (hips) | 88
  RLL> 2mm in all zones at 4 years | 0
  RLL> 2mm in all zones at 5 years: number analyzed (Participants) | 70
  RLL> 2mm in all zones at 5 years: number analyzed (hips) | 70
  RLL> 2mm in all zones at 5 years | 0

5. Secondary Outcome: Radiographic Outcomes: Migration of the Acetabular Shell Greater Than 5 mm in Any Direction
Description: Defined as the measurable change in the acetabular shell position relative to reproducible bony landmarks.
Time Frame: 3 month, 1, 2, 3, 4, 5 years
Population: Participants/hips are based on evaluable films for this data point. Overall number of participants and hips is based upon the 3 month population.
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | Trident® Tritanium™ Acetabular Shell
Number analyzed (Participants) | 156
Number analyzed (hips) | 158
hips
  Migration >5mm at 3 months | 0
  Migration >5mm at 1 year: number analyzed (Participants) | 137
  Migration >5mm at 1 year: number analyzed (hips) | 139
  Migration >5mm at 1 year | 0
  Migration >5mm at 2 years: number analyzed (Participants) | 123
  Migration >5mm at 2 years: number analyzed (hips) | 124
  Migration >5mm at 2 years | 0
  Migration >5mm at 3 years: number analyzed (Participants) | 95
  Migration >5mm at 3 years: number analyzed (hips) | 95
  Migration >5mm at 3 years | 0
  Migration >5mm at 4 years: number analyzed (Participants) | 90
  Migration >5mm at 4 years: number analyzed (hips) | 91
  Migration >5mm at 4 years | 0
  Migration >5mm at 5 years: number analyzed (Participants) | 73
  Migration >5mm at 5 years: number analyzed (hips) | 73
  Migration >5mm at 5 years | 0

6. Secondary Outcome: Change in Lower Extremity Activity Scale (LEAS) From Pre-operative to Post-operative
Description: The change in LEAS is reported by comparing the mean pre-operative, 3 month, 1, 2, 3, 4, and 5 year scores. The LEAS is completed by the participant to assess activity level. Activity levels were ordered in terms of intensity from 1 to 18, with 18 indicating the highest activity level.
Time Frame: pre-op, 3 month, 1, 2, 3, 4, 5 years
Population: Participants/hips with available data. Overall number of participants and hips analysed is based upon the preoperative population.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: hips
Arm/Group | Trident® Tritanium™ Acetabular Shell
Number analyzed (Participants) | 186
Number analyzed (hips) | 189
units on a scale
  LEAS preoperative | 8.32 (3.27)
  LEAS 3 month: number analyzed (Participants) | 163
  LEAS 3 month: number analyzed (hips) | 165
  LEAS 3 month | 9.25 (2.74)
  LEAS 1 year: number analyzed (Participants) | 145
  LEAS 1 year: number analyzed (hips) | 147
  LEAS 1 year | 10.5 (2.95)
  LEAS 2 years: number analyzed (Participants) | 123
  LEAS 2 years: number analyzed (hips) | 125
  LEAS 2 years | 10.37 (3.25)
  LEAS 3 years: number analyzed (Participants) | 105
  LEAS 3 years: number analyzed (hips) | 106
  LEAS 3 years | 10.6 (3.26)
  LEAS 4 years: number analyzed (Participants) | 100
  LEAS 4 years: number analyzed (hips) | 101
  LEAS 4 years | 10.25 (3.18)
  LEAS 5 years: number analyzed (Participants) | 84
  LEAS 5 years: number analyzed (hips) | 85
  LEAS 5 years | 10.15 (3.16)
Statistical Analysis 1: Comparison: Trident® Tritanium™ Acetabular Shell; Test type: Other — To test whether the change from the pre-operative LEAS Score compared to the 3 month LEAS Score is statistically significant; p = 0.0011, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: Trident® Tritanium™ Acetabular Shell; Test type: Other — To test whether the change from the pre-operative LEAS compared to the 1, 2 and 3 year LEAS are statistically significant; p < 0.0001, t-test, 2 sided — This p-value applies to pre-op to 1, 2 and 3 year intervals; Paired t-test
Statistical Analysis 3: Comparison: Trident® Tritanium™ Acetabular Shell; Test type: Other — To test whether the change from the pre-operative LEAS compared to the 4 year LEAS is statistically significant; p = 0.0002, t-test, 2 sided; Paired t-test
Statistical Analysis 4: Comparison: Trident® Tritanium™ Acetabular Shell; Test type: Other — To test whether the change from the pre-operative LEAS compared to the 5 year LEAS is statistically significant; p = 0.0009, t-test, 2 sided; Paired t-test

ADVERSE EVENTS:
Time Frame: Reportable adverse events for this study include those that are serious or related to the device.
Description: Censored protocol deviations were not included as at risk participants. Industry standard AE terms not used; specific AE terms not used for all AEs. Elective procedures not included. e.g.non-study joint replacement/revision, rotator cuff repair, carpal tunnel release, cataract, intra-ocular & bunion procedures, total shoulder repair, laminectomy, microdiscectomy, breast reduction, cervical spine fusion, & mid-foot/flat-foot surgery.
Groups:
- Operative Site Events: Trident® Tritanium™ Acetabular Shell used in revision total hip replacement. Operative site events are reported by hip.
- Non-operative Site Events: Trident® Tritanium™ Acetabular Shell used in revision total hip replacement. Non-Operative site events are reported by participant.
Arm/Group | Operative Site Events | Non-operative Site Events
Serious Adverse Events (participants affected / at risk) | 28/193 | 41/190
Other Adverse Events (participants affected / at risk) | 0/193 | 0/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Operative Site Events (N=193) | Non-operative Site Events (N=190)
Non-operative site (Cardiac disorders) | 0/0 (0) | 10 (11)
Non-operative site (Gastrointestinal disorders) | 0/0 (0) | 2 (3)
Non-operative site (General disorders) | 0/0 (0) | 6 (6)
Non-operative site (Hepatobiliary disorders) | 0/0 (0) | 1 (1)
Operative site (Infections and infestations) | 9 (10) | 0/0 (0)
Non-operative site (Infections and infestations) | 0/0 (0) | 9 (9)
Non-operative site (Metabolism and nutrition disorders) | 0/0 (0) | 2 (2)
Operative site (Musculoskeletal and connective tissue disorders) | 18 (19) | 0/0 (0)
Non-operative site (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 10 (10)
Non-operative site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 5 (7)
Non-operative site (Nervous system disorders) | 0/0 (0) | 1 (1)
Non-operative site (Renal and urinary disorders) | 0/0 (0) | 2 (2)
Non-operative site (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 2 (2)
Non-operative site (Vascular disorders) | 0/0 (0) | 5 (5)
Operative site (Vascular disorders) | 1 (1) | 0/0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each investigator shall have privileges for their own center's results at the completion of the study.These manuscripts & abstracts will be delayed until after the multi-center publication is submitted.All publications shall be submitted to the sponsor for review at least 60 days prior to the submission for publication.The sponsor shall not edit or otherwise influence the publications other than to ensure that confidential information is not disclosed and that the data is accurately represented.